CLINICAL TRIAL: NCT04599738
Title: The Effect of Millet-based Muffins on Glycaemic, Insulinemic Response and Gastric Emptying in Pre-diabetic Adults
Brief Title: Millet-based Muffins, Glycaemic Response, Insulinemic Response and Gastric Emptying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Collaborators: Taibah University (Other)
Responsible Party: Principal Investigator, Dr. Sangeetha Thondre, Senior Lecturer, Oxford Brookes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UREC 161061
Record Dates: First submitted 2020-10-11; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Healthy; Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wheat muffin (Placebo Comparator): Muffin made with 100% wheat flour
  Interventions: Other: Wheat muffin
- Finger millet grain muffin (Experimental): Muffin made with 50% wheat flour and 50% finger millet crushed grain
  Interventions: Other: Finger millet grain muffin

INTERVENTIONS:
Other: Wheat muffin — Participants consumed a control muffin made of wheat flour.
  Arms: Wheat muffin
Other: Finger millet grain muffin — Participants consumed a test muffin made of finger millet grain and wheat flour.
  Arms: Finger millet grain muffin

SUMMARY:
Millet is a functional grain that has attracted the attention of scientists for many years due to its significant benefits to human health. Research has shown that millets have a high antioxidant capacity and polyphenol content which can contribute to a reduced risk of some chronic diseases such as type 2 diabetes and its complications. This study aimed to assess the glycaemic response (GR), insulinaemic response (IR) and gastric emptying (GE) after the consumption of millet-based muffins in pre-diabetic and healthy participants.

This was a single-blind, randomized controlled crossover study in which participants consumed one control muffin (wheat) and one test muffin (millet). During each session, participants were required to consume either the test or the control muffin, consuming the alternative on the next visit. Then, 10 finger-prick blood samples were taken for the determination of glucose and insulin over 4 hours. 13Carbon (13C) sodium acetate was added to the muffins (control and test) in order to measure gastric emptying from the breath samples collected.

DETAILED DESCRIPTION:
This study aimed to assess the glycaemic response (GR), insulinaemic response (IR) and gastric emptying (GE) after the consumption of millet-based muffins in pre-diabetic and healthy participants. This was a single-blind, randomized controlled crossover study in which participants consumed one control muffin (wheat) and one test muffin (millet).This study investigated the effect of polyphenol-rich millet-based muffin on glycaemic response (GR), insulinaemic response (IR) and gastric emptying (GE) in healthy and pre-diabetic participants (people with prediabetes have blood glucose levels that are higher than normal but not yet high enough to be diagnosed as diabetes - the normal fasting blood glucose level is below 6.1 mmol/l or 108 mg/dl).

After potential participants have read the Participant Information Sheet (PIS) and signed the consent form, they were screened during the first visit to measure fasting blood glucose (FBG; fasting blood glucose should be between 6.1 to 6.9 mmol/l for pre-diabetic participants and < 6.1 mmol/l for healthy participants ).If eligible for the study, body weight and height and blood pressure were taken in the Functional Food Centre (currently known as Oxford Brookes Centre for Nutrition and Health). If the fasting blood glucose test was less than 6.1mmol/l (participants were informed of their fasting blood glucose result and given the choice either to do Oral glucose tolerance test (OGTT) to check for Impaired Glucose Tolerance (IGT), participate in the healthy group or to be excluded). If the participant agreed to continue and had one or more of the pre-diabetes inclusion criteria, they could complete an oral glucose tolerance test (OGTT) over 2 hours.( An oral glucose tolerance test involves taking a fasting sample of blood and then taking a very sweet drink containing 75g of glucose. After having this drink participants had to stay at rest until a further blood sample is taken after 2 hours.) If their 2 h blood glucose result was between 7.9 to 11.0 mmol/l, they were considered eligible to participate in the study as a prediabetic participant, and were asked to come for a subsequent visit in order to begin the study. If the participant does not have IGT, they had the option to take part in the study as a healthy participant.

ELIGIBILITY:
Inclusion Criteria:

* for healthy participants

  * Aged 18-65 years
  * Body mass index (BMI) ≤ 30kg/m2
  * Fasting blood glucose < 6.1 mmol/l
  * Non-pregnant and non-lactating
  * No known diabetes or impaired glucose tolerance
  * No medical condition(s) or medication(s) known to affect glucose regulation or appetite and/or which influence digestion and absorption of nutrients
  * No major medical or surgical event requiring hospitalisation within the preceding three months
  * No use of steroids, protease inhibitors or antipsychotics
  * No food allergy to millet, wheat, egg and milk.

At least one of the following for pre-diabetes participants Fasting blood glucose 6.1-6.9 mmol/l (108-125 mg/ dI) - (WHO, 2006) or/and an Oral glucose tolerance test (OGTT) at 2 hours 7.9 to 11.0 mmol/l

Exclusion Criteria:

* • Pregnant and lactating

  * Diabetes
  * Medical condition(s) or medication(s) known to affect glucose regulation or appetite and/or which influence digestion and absorption of nutrients
  * Medical or surgical event requiring hospitalisation within the preceding three months
  * Use of steroids, protease inhibitors or antipsychotics (because of their effects on glucose regulation of appetite or influence digestion and absorption of nutrients).
  * Food allergy to study products (millet. wheat, egg, milk, butter, sugar).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-12-24 (Actual); Study Completion 2017-12-24 (Actual)

PRIMARY OUTCOMES:
Change in glycaemic response from baseline for 180 minutes | 180 minutes
  Capillary blood glucose was measured for 180 minutes at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
Change in insulin response from baseline for 180 minutes | 180 minutes
  Capillary plasma insulin was measured for 180 minutes at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes

SECONDARY OUTCOMES:
Gastric emptying for 4 hours | 4 hours
  Breath samples were taken at every 15 minutes for 4 hours
Satiety by visual analogue scale for 4 hours | 4hours
  Visual analogues scale. The rating of the scale was: 6 = extremely full and 0 = extremely hungry. Higher score meant a better outcome of increased satiety.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Thondre, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes Centre for Nutrition and Health, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following registration
Access Criteria: Upon request

REFERENCES:
- [Background] Brouns F, Bjorck I, Frayn KN, Gibbs AL, Lang V, Slama G, Wolever TM. Glycaemic index methodology. Nutr Res Rev. 2005 Jun;18(1):145-71. doi: 10.1079/NRR2005100. PMID 19079901
- [Background] Carbohydrates in human nutrition. Report of a Joint FAO/WHO Expert Consultation. FAO Food Nutr Pap. 1998;66:1-140. No abstract available. PMID 9743703
- See also: Food Products-Determination of the glycaemic index (GI) and recommendation for food classification. — http://www.iso.org/standard/43633.html
- Available data/document: Study Protocol — https://drive.google.com/drive/u/0/folders/1wsl_6XU0myZgcXtOjRaemk414v9qgDaz
- Available data/document: Informed Consent Form — https://drive.google.com/drive/u/0/folders/1wsl_6XU0myZgcXtOjRaemk414v9qgDaz

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT04599738/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT04599738/ICF_001.pdf